CLINICAL TRIAL: NCT02891629
Title: Safety and Feasibility of the EyeControl Device (Eye-based Communication Device) for ALS Patients
Brief Title: Safety and Feasibility of the EyeControl Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eyefree Assisting Communication Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EFAC-01
Record Dates: First submitted 2016-08-29; First posted 2016-09-07 (Estimated); Results first posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: ALS (Amyotrophic Lateral Sclerosis)
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Device use in Healthy volunteers (Experimental): 10 healthy volunteers will be recruited
  Interventions: Device: EyeControl device
- Device use in ALS patients (Experimental): 5 ALS patients in early stages will be recruited
  Interventions: Device: EyeControl device

INTERVENTIONS:
Device: EyeControl device — Use of device features including control of gestures, use of menus, activation of pre- defined modes and writing full sentences

SUMMARY:
The EyeControl device is an eye movement-based communication device in the form of wearable glasses with connected infrared cam-era that tracks the pupil and translates blinks and movements into commands.This study is aimed to demonstrate the safety and feasibility of the EyeControl device in healthy volunteers, and ALS patients in early stages.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects 18 to 65 years old
2. Subject with understandable speaking communication
3. Subject fluent in Hebrew (speech and writing skills)

   Additional inclusion criteria for Stage 2 of the study:
4. Subjects with early stage ALS diagnosis - whose speech capability is unaffected

Exclusion Criteria:

1. Subjects with glasses or contact lenses
2. Subjects with eye conditions such as Ptosis, Strabismus And Crossed Eyes
3. Medical history of epilepsy
4. Subjects who according to investigator's judgement, unable to comply with the requirements of this protocol
5. Pregnant or lactating women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-01-28 (Actual); Study Completion 2017-02-28 (Actual)

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Investigator decided to terminate subject participation due to the discovery of cataract during the trial.
Period: Overall Study
Arm/Group | Device Use in Healthy Volunteers | Device Use in ALS Patients
Started | 10 | 5
Completed | 10 | 4
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Device Use in Healthy Volunteers | Device Use in ALS Patients | Total
Number analyzed (Participants) | 10 | 4 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 4 | 14
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.3 (9.83) | 46.25 (5.26) | 36.6 (11.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 0 | 5
  Male | 5 | 4 | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Israel | 10 | 4 | 14

OUTCOME MEASURES:

1. Primary Outcome: Feasibility - Successful Performance Rate of Device Features
Description: Ability to successfully perform at least 70% of device features (controlling the application and Free text features)
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Device Use in Healthy Volunteers | Device Use in ALS Patients
Number analyzed (Participants) | 10 | 4
seconds | 4.9 (1.3) | 7.2 (2.2)

2. Secondary Outcome: Safety Assessment - Number of Device Related Adverse Events
Description: number of device related adverse events reported during the use of the device
Time Frame: 2 weeks
Measure: Number; unit: events
Arm/Group | Device Use in Healthy Volunteers | Device Use in ALS Patients
Number analyzed (Participants) | 10 | 4
events | 2 | 0

ADVERSE EVENTS:
Time Frame: The adverse events data was collected only during the trial, meaning during the 4 sessions, of about 2.5-3 hours, for each participant, performed over 2 weeks' time.
Description: An AE can be any unintended sign, symptom, disease or injury or any untoward clinical signs (including an abnormal laboratory findings) in subjects, users or other persons whether or not related to the investigational medical device.
Arm/Group | Device Use in Healthy Volunteers | Device Use in ALS Patients
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/5
Other Adverse Events (participants affected / at risk) | 1/10 | 0/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Device Use in Healthy Volunteers (N=10) | Device Use in ALS Patients (N=5)
Dry Eyes (Eye disorders) | 1 (1) | NA — Participant complained on dry eyes
Eye Fatigue (Eye disorders) | 1 (1) | NA — Participant complained on eye fatigue

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2016-05-16): https://cdn.clinicaltrials.gov/large-docs/29/NCT02891629/Prot_000.pdf